CLINICAL TRIAL: NCT03690115
Title: Phase 2 Study of Ponatinib (Iclusig) for Prevention of Relapse After Allogeneic Stem Cell Transplantation (allo-SCT) in FLT3-ITD AML Patients: the PONALLO Trial."
Brief Title: Study of Ponatinib (Iclusig) for Prevention of Relapse After Allogeneic Stem Cell Transplantation (allo-SCT) in FLT3-ITD AML Patients
Acronym: PONALLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Patrice Chevallier, investigator coordinator, Nantes University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1701_ PONALLO
Record Dates: First submitted 2018-04-04; First posted 2018-10-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Administration of ponatinib after allo-SCT transplant in FLT3-ITD AML patient
  Interventions: Drug: Ponatinib 30 MG

INTERVENTIONS:
Drug: Ponatinib 30 MG — Administration of ponatinib after allo-SCT transplant in FLT3-ITD AML patient

SUMMARY:
Recent advances in acute myeloid leukemia (AML) have been characterized by a better understanding of disease biology. As such, FMS-like tyrosine kinase 3-internal tandem duplication (FLT3-ITD) have been recognized as conferring a poor prognosis. The FLT3-ITD molecular mutation is observed in about one-quarter of patients diagnosed with AML. Patients presenting with this abnormality are referred for early allogeneic stem-cell transplantation (allo-SCT). However, some data suggest that FLT3-ITD remains associated with a poor prognosis even after allo-SCT because of higher risk of relapse and strategies for preventing relapse in the post-transplant setting are required (Hu et al, Expert Rev Hematol, 2014). For example, in a large cohort of patients (Brunet et al, JCO, 2012), the incidence of relapse for FLT3-ITD AML patients after allo-SCT was 30% at 2-years, significantly higher compared to FLT3-ITD negative patients (p=0.006).

Ponatinib (Iclusig®) is an orally available, tyrosine kinase inhibitor with a unique binding mechanism allowing inhibition of BCR-ABL kinases, including those with the T315I point mutation. Ponatinib also has in vitro inhibitory activity against a discrete set of kinases implicated in the pathogenesis of other hematologic malignancies, including FLT3, KIT, fibroblast growth factor receptor 1 (FGFR1), and platelet derived growth factor receptor α (PDGFRα). In vitro activity of ponatinib in AML has been already demonstrated (Gozgit et al, Mol Cancer Ther, 2011; Smith et al, Blood 2013). If some trials are on-going to test ponatinib alone or in combination with chemotherapy in FLT3-ITD AML (Clinical.trials.gov), no study is dedicated to the use of ponatinib in the post-transplant setting in order to prevent relapse in these patients.

The main goal of this study will be to determine the maximal tolerated dose (MDT) of ponatinib after allo-SCT in FLT3-ITD AML patients, then to investigate the efficacy of ponatinib in a larger cohort of patients

ELIGIBILITY:
Inclusion Criteria:

* Engraftment
* Controlled GVHD
* Positive FLT-3 ITD AML in cytologic complete remission
* Have an Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Have adequate renal function: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) for institution
* Have adequate hepatic function: Total serum bilirubin ≤ 1.5 × ULN, unless due to Gilbert's syndrome; Alanine aminotransferase (ALT) ≤ 2.5 × ULN, or ≤ 5 × ULN if leukemic infiltration of the liver is present ; Aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5 × ULN if leukemic infiltration of the liver is present
* Have normal pancreatic status: Serum lipase and amylase ≤ 1.5 × ULN
* Have normal QTcF interval on screening electrocardiogram (ECG) evaluation,defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
* Platelets ≥ 100 Giga/l; Neutrophils ≥ 1 Giga/l
* Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
* Agree to use an effective form of contraception with sexual partners throughout study participation (for female and male patients who are fertile).
* Provide written informed consent.
* Be willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

* HIV positive, active Hepatitis B or C
* Childbearing or childbreast feeding women
* Women or men without effective contraceptive barrier if needed
* Previous myocardial infarction, or cerebral vascular accident, pancreatitis
* Respiratory insufficiency defined as DLCO <40% of the corrected value
* Creatinine clearance ≤ 50ml/min
* Contra-indication to ponatinib
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Patients at high or very high risk of cardiovascular disease with any of the following

  1. Established cardiovascular disease Cardiac disease:

     * Congestive heart failure greater than class II NYHA or
     * Left ventricular ejection fraction (LVEF) < 50% or
     * Unstable angina (anginal symptoms at rest) or
     * New onset angina (began within the last 3 months) or
     * Myocardial infarction, coronary/peripheral artery disease, congestive heart failure, cerebrovascular accident including transient ischemic attack within the past 12 months or
     * History of thrombolic or embolic events Arrhythmias
     * Any history of clinically significant cardiac arrhythmias requiring anti-arrhythmic therapy.
  2. Diabetes Mellitus,
  3. Arterial Hypertension,

     * Uncontrolled hypertension defined as systolic blood pressure greater than 140 mmHg or diastolic pressure greater than 90 mmHg, despite optimal medical management and optimal measurement (http://www.has-sante.fr/portail/display.jsp?id=c_272459)
     * Any history of hypertension with
     * Hypertensive encephalopathy
     * Posterior leucoencephalopathy
     * Aortic or artery dissection
  4. Familial dysplipidemia.
  5. Taking medications that are known to be associated with Torsades de Pointes (see

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Relapse incidence at 2 years from transplant | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
  time interval from the graft (day 0) until the date of last follow-up or death
Leukemia free survival | 2 years
  time interval from the date of the graft (day 0) until the date of last follow-up, death or relapse
Non-relapse mortality (NRM) | day 100
  incidence of mortality due to all causes except relapse after transplant, considering that cause of death for patients having relapsed but dying from another cause is relapse
Acute and chronic GVHD | 2 years
  NIH score
Influence of Ponatinib on Immune reconstitution PB lymphocyte cells | 1 years
  an immunophenotype of PB lymphocytes will be performed by flow cytometry at +3, +6, +9 and +12 months post-transplant to study the reconstitutions of CD3, CD4 and CD8 T cells, B and NK cells. The results will be expressed as absolute counts (Giga/L). We want to establish the potential influence of ponatinib on the reconstitution of these cells
Inflence of Ponatinib on Chimerism of Donor peripheral blood and CD3 T cells | 1 years
  Donor peripheral blood and CD3 T cells chimerism will be studied using molecular markers and RT-PCR at day +30, +60, +90, and +6, +12 months post-transplant. We want to establish the potential influence of ponatinib on the chimerism post-transplant.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Angers, Angers
  - CHu Brest, Brest
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Chevallier, Nantes
  - Hopital St Antoine, Paris
  - Hopital St Louis, Paris
  - CHu Lyon, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CRLC Toulouse, Toulouse
  - CHU Nancy, Vandœuvre-lès-Nancy